CLINICAL TRIAL: NCT02032914
Title: The Prevalence of Colonic Neoplasm in Cryptogenic Pyogenic Liver Abscess
Brief Title: Prevalence of Colon Cancer in Pyogenic Liver Abscess
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Tae Oh Kim, Assistant professor, Inje University
Other Study IDs: 1
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Cryptogenic Pyogenic Liver Abscess
Keywords: pyogenic liver abscess; colon cancer
MeSH Terms: conditions — Liver Abscess, Pyogenic; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonoscopic examination group: The patients diagnosed with cryptogenic pyogenic liver abscess

SUMMARY:
Although a proportion of pyogenic liver abscess may originated from colonic mucosal lesions, the prevalence of colonic neoplasm in the patients with pyogenic liver abscess are still not evaluated yet. Thus, our group will find the prevalence of colonic neoplasm in the group of cryptogenic pyogenic liver abscess by colonoscopic examination.

ELIGIBILITY:
Inclusion Criteria:

* Pyogenic liver abscess radiologically and bacteriologically diagnosed

Exclusion Criteria:

* Amebic liver abscess
* Other causes of pyogenic liver abscess such as cholangitis, liver cancer, complication of transarterial chemoembolization or radiofrequency ablation to hepatocellular carcinoma
* Refusal to colonoscopic examination
* Inadequate general patient status to perform the colonoscopic examination
* Patient who has had the screening colonoscopic examination within 1 year and showed normal finding or had 1 or 2 colon polyp in adequate exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients diagnosed as pyogenic liver abscess, the cause of which is not found at initial evaluation
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The prevalence of colonic neoplasm | within 6 weeks after diagnosis of pyogenic liver abscess

SECONDARY OUTCOMES:
Prevalence of colon polyp | Within 6 weeks at diagnosis of pyogenic liver abscess
Prevalence of colonic diverticulitis | Within 6 weeks at diagnosis of pyogenic liver abscess
Prevalence of inflammatory bowel disease | Within 6 weeks at diagnosis of pyogenic liver abscess
Prevalence of intestinal tuberculosis | Within 6 weeks at diagnosis of pyogenic liver abscess

CONTACTS AND LOCATIONS:
Overall Officials: Tae Oh Kim, M.D., Principal Investigator — Inje University Haeundae Paik Hosptial
Locations (2):
- South Korea (2):
  - Pusan National Unversity Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Inje University Haeundae Paik Hospital, Busan